CLINICAL TRIAL: NCT03299439
Title: A Multi-center Randomized Controlled Trial of Acupuncture Treatment for Knee Osteoarthritis With Sensitive Acupoints and Tender Points
Brief Title: Acupuncture Treatment for Knee Osteoarthritis With Sensitive Acupoints and Tender Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Sun Xin, Director, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20178159950025
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Acupuncture; Knee Osteoarthritis; Sensitive Acupoints; Tender Points
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acupuncture at highly sensitive points (Experimental): Sterile, single-use filiform acupuncture needles (Hwato Needles, Sino-foreign Joint Venture Suzhou Hwato Medical Instruments Co., China) with a length of 40 mm and a diameter of 0.30 mm will be inserted to a depth of 15-30mm in five highly sensitive points.
  Interventions: Other: acupuncture
- acupuncture at lowly/non-sensitive points (Active Comparator): Sterile, single-use filiform acupuncture needles (Hwato Needles, Sino-foreign Joint Venture Suzhou Hwato Medical Instruments Co., China) with a length of 40 mm and a diameter of 0.30 mm will be inserted to a depth of 15-30mm in five low/non-sensitive points.
  Interventions: Other: acupuncture
- no acupuncture (waiting-list) (No Intervention): Patients in the waiting-list group will not receive any acupuncture intervention during the study.

INTERVENTIONS:
Other: acupuncture — a stimulation of the body or auricular points
  Arms: acupuncture at highly sensitive points; acupuncture at lowly/non-sensitive points

SUMMARY:
The investigators plan to investigate the effectiveness of acupuncture at highly sensitive points, compared with lowly/non-sensitive points or no acupuncture (waiting-list), in improving pain, joint function and quality of life, among patients with KOA. The safety of acupuncture will also be assessed during the study period.

DETAILED DESCRIPTION:
Participants in the high sensitization group receive acupuncture treatment at the five highly sensitive points; Participants in the low/non-sensitization group receive acupuncture treatment at the five low/non-sensitive points and all other treatment settings will be the same as in the high sensitization group. Patients in the waiting-list group will receive standard acupuncture treatment after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 40 years or older and diagnosed with mild or moderate knee osteoarthritis(KOA) are eligible to participate in the study
* The following criteria are used for diagnosis of KOA:

  * refractory knee pain for most days in the last month;
  * joint space narrowing, sclerosis or cystic change in subchondral bone (as demonstrated in X-ray);
  * laboratory examinations of arthritis: clear and viscous synovial fluid (≥2 times) and white blood cell count < 2000/mm3;
  * morning stiffness continues less than 30 minutes;
  * bone sound exists when joints was taking flexion and/or extension. If a patient meets criteria 1 and 2, or criteria 1, 3, 4, and 5, a diagnosis of KOA is confirmed.

Exclusion Criteria:

Patients will be excluded if they meet any of the following:

* diagnosed with conditions leading to skeletal disorders, such as tuberculosis, tumors or rheumatism of the knee joint and rheumatoid arthritis;
* present sprain or trauma in the lower limb;
* unable to walk properly due to foot deformity or pain;
* present with mental disorders;
* present with comorbidities including severe cardiovascular disease, liver or kidney impairment, immunodeficiency, diabetes mellitus, blood disorder or skin disease;
* females who are pregnant or lactating;
* using physiotherapy treatments for osteoarthritis knee pain;
* have used intra-articular injection of glucocorticoid or viscosupplementation in the past six months;
* received knee-replacement surgery;
* diagnosed with severe (stage 4, according to Kellgren and Lawrence radiographic classification) or late clinical stage of KOA;
* have a swollen knee or positive result of floating patella test; or'
* are participating or have participated in the other clinical trials.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
The change of Western Ontario and McMaster Universities Osteoarthritis index total score from baseline to 16 weeks | Assessments will be conducted at baseline and 16 weeks after randomization
  It consists of 24 items assessing the knee osteoarthritis patients pain, stiffness, and physical function. Each of the 24 items will be graded on a visual analog scale ranging from 0 to 10, with higher scores reflecting more pain, stiffness and poorer physical function.

SECONDARY OUTCOMES:
The change of Short Form (SF)-12 health survey score from baseline to 16 weeks | Assessments will be conducted at baseline and 16 weeks after randomization
  It includes 12 items: 2 items on physical functioning, 2 items on role limitations because of physical health problems, 1 item on bodily pain, 1 item on general health perceptions, 1 item on vitality (energy/fatigue), 1 item on social functioning, 2 items on role limitations because of emotional problems, and 2 items on general mental health (psychological distress and psychological well-being).
The changes of knee ranges of motion (ROMs) from baseline to 16 weeks | Assessments will be conducted at baseline and 16 weeks after randomization
  The knee ROMs will be assessed both actively and passively by using a standard goniometer. It will include flexion, extension, internal rotation and external rotation.
The changes of pressure-pain threshold of the five selected acupuncture points from baseline to 16 weeks | Assessments will be conducted at baseline and 16 weeks after randomization
  The pressure-pain threshold of the five selected acupuncture points will be measured using the electronic von Frey detector.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, Phd, Study Chair — West China Hospital
Locations (4):
- China (4):
  - the Third Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan
  - Wuhan Integrated Traditional Chinese Medicine and Western Medicine Hospital, Wuhan, Hubei
  - Department of Integrated Traditional Chinese and Western Medicine, West China Hospital, Sichuan University, Chengdu, Sichuan
  - the Affiliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu J, Li Y, Li L, Luo X, Li N, Yang X, Zhang H, Liu Z, Kang D, Luo Y, Liu Y, Jia Y, Ren Y, Yao M, Wang Y, Chen J, Maiji M, Zou K, Zhao L, Liang F, Sun X. Effects of acupuncture at acupoints with lower versus higher pain threshold for knee osteoarthritis: a multicenter randomized controlled trial. Chin Med. 2022 Jun 8;17(1):67. doi: 10.1186/s13020-022-00626-3. PMID 35676697
- [Derived] Tang L, Jia P, Zhao L, Kang D, Luo Y, Liu J, Li L, Zheng H, Li Y, Li N, Guyatt G, Sun X. Acupuncture treatment for knee osteoarthritis with sensitive points: protocol for a multicentre randomised controlled trial. BMJ Open. 2018 Oct 2;8(10):e023838. doi: 10.1136/bmjopen-2018-023838. PMID 30282686

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT03299439/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT03299439/ICF_001.pdf